CLINICAL TRIAL: NCT05620732
Title: Efficacy and Safety of Claudin18.2CAR-T in Advanced Pancreatic Cancer and Gastric Carcinoma
Brief Title: Treatment of Advanced Malignant Solid Tumors With Claudin18.2CAR-T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-025
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Advanced Pancreatic Carcinoma; Advanced Gastric Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients treated with Claudin 18.2 CAR-T cells.
  Interventions: Biological: Claudin18.2 CAR-T cells

INTERVENTIONS:
Biological: Claudin18.2 CAR-T cells — patients treated with Claudin18.2 CAR-T cells

SUMMARY:
The efficacy of advanced pancreatic cancer and gastric cancer needs to be further improved. Claudin is a kind of integrin membrane protein in the tight junction between epithelium and endothelium, which is highly expressed in gastric cancer and pancreatic cancer. Preclinical studies suggest that Claudin18.2CAR-T can effectively improve the remission rate of patients with advanced solid tumors.

DETAILED DESCRIPTION:
The efficacy of advanced pancreatic cancer and gastric cancer needs to be further improved.

Claudin is a kind of integrin membrane protein in the tight junction between epithelium and endothelium, which is highly expressed in gastric cancer and pancreatic cancer. Preclinical studies suggest that Claudin18.2CAR-T can effectively improve the remission rate of patients with advanced solid tumors.

Investigators aim to testify to the safety and efficacy of Claudin18.2CAR-T cells in advanced pancreatic cancer and gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (≥ 18, ≤ 75), regardless of gender;
2. Subjects voluntarily participate in the study, and they or their legal guardians sign the Informed Consent Form;
3. Non resectable, locally late recurrent or metastatic gastric cancer or pancreatic cancer confirmed by histopathology; Patients with gastric cancer or pancreatic cancer diagnosed as stage III or IV according to the TNM staging system of the American Joint Commission on Cancer (AJCC) (8th edition in 2017);
4. According to RECIST 1.1 standard, there are clearly measurable and evaluable lesions;
5. Immunohistochemical staining confirmed that Claudin 18.2 was moderately and highly expressed in tumor tissues;
6. Subjects must have received the first and second line standard treatment scheme;
7. The subject must not be suitable for receiving radical treatment methods, such as radical chemotherapy and radiotherapy and/or surgery/immunosuppressant at the checkpoint, or refuse surgical resection
8. Within 2 weeks before cell therapy, no antibody drugs were used;
9. ECOG score is 0-2;
10. The subjects had no contraindication for peripheral blood collection;
11. The expected survival period is more than 3 months.

Exclusion Criteria:

1. People who have a history of allergy to any component in cell products;
2. The following conditions occur in blood routine examination: WBC ≤ 1 × 109/L, absolute value of central granulocyte ANC ≤ 0.5 × 109/L, absolute value of lymphocyte ALC ≤ 0.5 × 109/L , PLT≦25 × 109/L ；
3. The following conditions occur in laboratory testing: including but not limited to, total serum bilirubin ≥ 1.5mg/dl; Serum ALT or AST is more than 2.5 times of the upper limit of normal; Blood creatinine ≥ 2.0mg/dl;
4. According to the NYHA cardiac function grading standard, patients with cardiac insufficiency belong to Grade III or IV; Or left ventricular ejection fraction (LVEF)<50% by echocardiography;
5. Pulmonary function is abnormal, and the saturation of blood oxygen under indoor air is less than 92%;
6. Myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, or other serious heart diseases clinically within 12 months before enrollment;
7. Grade 3 hypertension and poor blood pressure control after drug treatment;
8. Have suffered from brain trauma, consciousness disorder, epilepsy, relatively serious cerebral ischemia or cerebral hemorrhage disease in the past;
9. Patients with autoimmune diseases, immunodeficiency or other patients requiring immunosuppressive treatment;
10. There is uncontrolled active infection;
11. Have used any CAR-T cell product or other genetically modified T cell therapy before;
12. Live vaccine inoculation within 4 weeks before enrollment;
13. HIV, HBV, HCV and TPPA/RPR positive persons, and HBV carriers;
14. Subjects have a history of alcohol abuse, drug abuse or mental illness;
15. Subjects have participated in any other clinical research within 3 months before joining this clinical research;
16. Female subjects have any of the following conditions: a) are in pregnancy/lactation; Or b) having a pregnancy plan during the trial; Or c) is fertile and unable to take effective contraceptive measures;
17. The investigator believes that there are other circumstances that are not suitable for the subject to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
AE/SAE | From date of infusion to 30 days after infusion
  adverse events/ severe adverse events

SECONDARY OUTCOMES:
ORR | From admission to the end of follow up, up to 2 years.
  overall response rate

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Dr, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Li Yu, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No